CLINICAL TRIAL: NCT04920526
Title: Effectiveness of the QHPV Among Kenyan HIV Infected Girls and Boys 9 Years Post Vaccination
Brief Title: Effectiveness and B-memory Cell Response to QHPV Vaccine 9-years Post-vaccination Among HIV-infected Boys and Girls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Nelly Rwamba Mugo, Principal Investigator, Kenya Medical Research Institute
Other Study IDs: MISP 60583
Record Dates: First submitted 2021-05-17; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: HPV-Related Carcinoma
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- QHPV Vaccine: all participants have received QHPV
  Interventions: Drug: Quadrivalent HPV [Type 6, 11, 16 and 18] L1 Virus-Like Particle Vaccine

INTERVENTIONS:
Drug: Quadrivalent HPV [Type 6, 11, 16 and 18] L1 Virus-Like Particle Vaccine — No intervention will be administered
  Other Names: Gardasil

SUMMARY:
In 2013, the Investigators enrolled a cohort of 180 HIV-1 infected adolescent girls and boys ages 9-14 years and administered three doses of the QHPV vaccine (NCT04711265). For this study, the Investigators shall evaluate vaccine effectiveness 9 years post first vaccination.

Participants will be evaluated for HPV type specific antibody, genital HPV infection, genital warts and a subset of 30 participants will be evaluated for memory B and T cell responses.

DETAILED DESCRIPTION:
Genital Human Papilloma Virus (HPV) infections occur rapidly after sexual debut, and immunosuppressed individuals are at greater risk for incident and persistent infection. HPV vaccine contains virus-like participles (VLP), which are highly immunogenic and induce a robust humoral response that has been demonstrated to confer long term protection from HPV infection and associated disease among HIV-uninfected individuals.

The magnitude of type-specific vaccine induced neutralizing HPV antibody responses are diminished among HIV-infected compared to uninfected individuals.

There is no established minimum level of antibody that predicts protection against HPV infection or associated disease, the impact of lower antibody titers among HIV infected individuals on vaccine efficacy is unknown. The risk of HPV exposure persists throughout a person's sexual life and the duration of protection, especially when the vaccine is given in the early adolescent period is critical to vaccine effectiveness. Long lasting memory is characterized by memory B cells and long-lived plasma cells and a QHPV booster dose has demonstrated an anamnestic response among HIV-infected adolescents.

HPV efficacy and effectiveness data for HIV-uninfected individuals has informed the current World Health Organization (WHO) two-dose vaccine schedule. The field lacks data on effectiveness of three dose or two-dose for the HIV-infected adolescents. The current on-going research for single dose schedules gives urgency to the determination of long-term efficacy of three HPV vaccine doses for the HIV-infected adolescent.

The Investigators shall recall HIV-infected girls and boys who were previously vaccinated at ages 9-14 years with three doses of the quadrivalent vaccine (QHPV) in 2014 and evaluated for vaccine immunogenicity.

Method: The participants will be assessed for genital warts and genital HPV infection. Type specific HPV DNA will be assessed using genital swabs and genital warts assessed through physical examination among sexually active participants at enrollment, month 6 &12.

A sub-set of study participants will receive a booster dose of QHPV and evaluated for memory B and T cell responses.

The total duration of study follow up will be 12 months

ELIGIBILITY:
Inclusion Criteria:

1. received three doses of the quadrivalent HPV vaccine and enrolled in the quadrivalent HPV vaccine safety and immunogenicity study (MISP 38406)
2. participant consent or parental/guardian consent and participant assent for participants still <18 years of age
3. participants and guardians who consented to be contacted for further evaluation and participation in research and
4. are willing to continue longer-term follow up.

Exclusion Criteria:

1. Did not participate in the quadrivalent HPV vaccine safety and immunogenicity study (MISP 38406)
2. Not willing or able to provide written informed consent/assent to participate in the study

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study aims to enroll 135 HIV-1 infected boys and girls, who previously received three doses of quadrivalent HPV vaccine in the safety and immunogenicity study (MISP 38406)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in persistent Genital HPV infection | The changes will be measured at baseline (enrolment), month 6 and 12
  Type specific HPV serotype: -6, -11, -16 and -18 and additional 13 oncogenic HPV serotypes 31,33,35,39,45,51,52,56,58,59,66, 68,73 as per International Agency for Research on Cancer (IARC) monographs.
Changes in geometric titers for HPV-specific Antibodies | This outcome will be measured at Month 12
  Vaccine type specific HPV antibody Geometric Mean Titers: HPV- 6, 11, 16 & 18
B-memory cell elicitation in the participants given a booster vaccine | This will be measured at 12 months after receiving a booster vaccine
  Elicited from Peripheral Blood Mononuclear Cell (PBMC)

CONTACTS AND LOCATIONS:
Overall Officials: Nelly R. Mugo, MMed Obs Gyn, Principal Investigator — University of Washington

REFERENCES:
- [Result] MacIntyre CR, Shaw P, Mackie FE, Boros C, Marshall H, Barnes M, Seale H, Kennedy SE, Moa A, Hayen A, Chughtai AA, O'Loughlin EV, Stormon M. Immunogenicity and persistence of immunity of a quadrivalent Human Papillomavirus (HPV) vaccine in immunocompromised children. Vaccine. 2016 Aug 5;34(36):4343-50. doi: 10.1016/j.vaccine.2016.06.049. Epub 2016 Jul 9. PMID 27406936
- [Result] Lehtinen M, Lagheden C, Luostarinen T, Eriksson T, Apter D, Harjula K, Kuortti M, Natunen K, Palmroth J, Petaja T, Pukkala E, Siitari-Mattila M, Struyf F, Nieminen P, Paavonen J, Dubin G, Dillner J. Ten-year follow-up of human papillomavirus vaccine efficacy against the most stringent cervical neoplasia end-point-registry-based follow-up of three cohorts from randomized trials. BMJ Open. 2017 Aug 18;7(8):e015867. doi: 10.1136/bmjopen-2017-015867. PMID 28821519
- [Result] Moscicki AB, Karalius B, Tassiopoulos K, Yao TJ, Jacobson DL, Patel K, Purswani M, Seage GR; Pediatric HIV/AIDS Cohort Study. Human Papillomavirus Antibody Levels and Quadrivalent Vaccine Clinical Effectiveness in Perinatally Human Immunodeficiency Virus-infected and Exposed, Uninfected Youth. Clin Infect Dis. 2019 Sep 13;69(7):1183-1191. doi: 10.1093/cid/ciy1040. PMID 30927547
- [Result] MacIntyre CR, Shaw PJ, Mackie FE, Boros C, Marshall H, Seale H, Kennedy SE, Moa A, Chughtai AA, Trent M, O'Loughlin EV, Stormon M. Long term follow up of persistence of immunity following quadrivalent Human Papillomavirus (HPV) vaccine in immunocompromised children. Vaccine. 2019 Sep 3;37(37):5630-5636. doi: 10.1016/j.vaccine.2019.07.072. Epub 2019 Aug 8. PMID 31402238
- [Result] Weinberg A, Huang S, Moscicki AB, Saah A, Levin MJ; IMPAACT P1085 Protocol Team. Persistence of memory B-cell and T-cell responses to the quadrivalent HPV vaccine in HIV-infected children. AIDS. 2018 Apr 24;32(7):851-860. doi: 10.1097/QAD.0000000000001773. PMID 29424778
- [Result] Einstein MH, Levin MJ, Chatterjee A, Chakhtoura N, Takacs P, Catteau G, Dessy FJ, Moris P, Lin L, Struyf F, Dubin G; HPV-010 Study Group. Comparative humoral and cellular immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and HPV-6/11/16/18 vaccine in healthy women aged 18-45 years: follow-up through Month 48 in a Phase III randomized study. Hum Vaccin Immunother. 2014;10(12):3455-65. doi: 10.4161/hv.36117. PMID 25483700
- [Result] Banatvala J, Van Damme P, Van Hattum J. Boosters for hepatitis B. European Consensus Group on Hepatitis B Immunity. Lancet. 2000 Jul 22;356(9226):337-8. doi: 10.1016/s0140-6736(05)73618-7. No abstract available. PMID 11071210
- [Result] Mugo NR, Eckert L, Magaret AS, Cheng A, Mwaniki L, Ngure K, Celum C, Baeten JM, Galloway DA, Wamalwa D, Wald A. Quadrivalent HPV vaccine in HIV-1-infected early adolescent girls and boys in Kenya: Month 7 and 12 post vaccine immunogenicity and correlation with immune status. Vaccine. 2018 Nov 12;36(46):7025-7032. doi: 10.1016/j.vaccine.2018.09.059. Epub 2018 Oct 5. PMID 30297124
- [Result] Pinto LA, Dillner J, Beddows S, Unger ER. Immunogenicity of HPV prophylactic vaccines: Serology assays and their use in HPV vaccine evaluation and development. Vaccine. 2018 Aug 6;36(32 Pt A):4792-4799. doi: 10.1016/j.vaccine.2017.11.089. Epub 2018 Feb 1. PMID 29361344
- [Result] Levin MJ, Huang S, Moscicki AB, Song LY, Read JS, Meyer WA, Saah AJ, Richardson K, Weinberg A; IMPAACT P1085 Protocol Team. Four-year persistence of type-specific immunity after quadrivalent human papillomavirus vaccination in HIV-infected children: Effect of a fourth dose of vaccine. Vaccine. 2017 Mar 23;35(13):1712-1720. doi: 10.1016/j.vaccine.2017.02.021. Epub 2017 Feb 24. PMID 28238631
- [Result] Pathak N, Dodds J, Zamora J, Khan K. Accuracy of urinary human papillomavirus testing for presence of cervical HPV: systematic review and meta-analysis. BMJ. 2014 Sep 16;349:g5264. doi: 10.1136/bmj.g5264. PMID 25232064
- [Result] Van Keer S, Tjalma WAA, Pattyn J, Biesmans S, Pieters Z, Van Ostade X, Ieven M, Van Damme P, Vorsters A. Human papillomavirus genotype and viral load agreement between paired first-void urine and clinician-collected cervical samples. Eur J Clin Microbiol Infect Dis. 2018 May;37(5):859-869. doi: 10.1007/s10096-017-3179-1. Epub 2018 Feb 7. PMID 29417310
- [Result] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Result] Smith JS, Lindsay L, Hoots B, Keys J, Franceschi S, Winer R, Clifford GM. Human papillomavirus type distribution in invasive cervical cancer and high-grade cervical lesions: a meta-analysis update. Int J Cancer. 2007 Aug 1;121(3):621-32. doi: 10.1002/ijc.22527. PMID 17405118
- See also: Gardasil product information — http://www.ema.europa.eu/en/documents/product-information/gardasil-9-epar-product-information_en.pdf